CLINICAL TRIAL: NCT00733850
Title: A Randomized, Open-Label, Safety and Exploratory Efficacy Study of Kanglaite Injection Plus Gemcitabine (G+K) Versus Gemcitabine in Patients With Advanced Pancreatic Cancer
Brief Title: Safety and Exploratory Efficacy of Kanglaite Injection in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KangLaiTe USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLT-PANC-001
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — kang-lai-te; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Kanglaite Injection plus Gemcitabine
  Interventions: Drug: Kanglaite Injection plus gemcitabine
- 2 (Active Comparator): Gemcitabine
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Kanglaite Injection plus gemcitabine — Intravenous repeating dose
  Other Names: KLT
  Arms: 1
Drug: Gemcitabine — Intravenous repeating dose
  Other Names: Gemzar
  Arms: 2

SUMMARY:
Gemcitabine is usually used to treat cancer of the pancreas. The purpose of this study is to determine if Kanglaite Injection (KLT) is safe in patients with cancer of the pancreas, and whether it improves the effectiveness of gemcitabine. Additionally, the effect, if any, of KLT on the signs and symptoms of cancer as well as the common side effects of chemotherapy will be evaluated.

The research drug, KLT, is purified from a traditional Chinese medicine called coix seed. It is approved in China for use in combination with chemotherapy to treat patients with advanced lung cancer and liver cancer. It is also approved in China for use by itself to treat the symptoms of cancer in patients with advanced cancer of any kind. In the US, KLT is purely experimental and is not approved for any use. While a small number of cancer patients in the US have received KLT alone in a Phase I study, this is the first US protocol to evaluate whether or not KLT is useful in pancreatic cancer.

This phase II clinical study was completed in the US in June 2014. The clinical study report was submitted to the FDA in January 2015. The designs of the phase III clinical study for KLT has been cleared by the FDA in May 2015 and will be launched soon.

ELIGIBILITY:
Inclusion Criteria:

* Must have a life expectancy of at least 84 days (12 weeks)
* Must be ambulatory and have either a Karnofsky performance status of 60 or higher or ECOG performance status of 0, 1 or 2
* Must have histologically confirmed pancreatic cancer, either locally invasive or metastatic, and not amenable to potentially curative resection
* Must have measurable or evaluable target lesions, by RECIST 1.1 criteria
* Must not have previously received chemotherapy for metastatic disease
* If female, must have negative pregnancy test, be at least one year post menopausal, or have undergone surgical sterilization and must be willing to use appropriate birth control measures unless post menopausal or post surgical sterilization
* Must be judged by the Investigator to have the initiative and means to be compliant with the protocol including the return for follow-up visits on schedule
* Must give written informed consent prior to any testing under this protocol
* Must have Hemoglobin > 9 gm/dl, WBC>2 x109/ml, and platelets >100,000/ul
* Must have Alkaline Phosphatase < 2.5 x ULN, ALT < 2.0 x ULN, AST< 2.0 x ULN and bilirubin < 2.0
* Must have stable renal function appropriate for age. A patient must have a serum creatinine of < 1.5mg/dl or a GFR > 60 mL/minute
* Must have a central venous catheter if randomized to the G + K arm of study, or if the patient does not have one, must agree to have one placed if randomized to the G+K arm.

Exclusion Criteria:

* Patient has a history of cancer within 5 years other than pancreatic cancer (excluding resected non melanoma skin carcinoma
* Patient has active (untreated or still receiving corticosteroids) brain metastases
* Patient has had prior chemotherapy for metastatic disease
* Patient has received prior gemcitabine < 12 months previously
* Patient is currently taking a bile acid sequestrant drug (such as Questran, Colestid or Welchol) or a fibric acid derivative drug (such as Lopid, Tricor, Antara, Lofibra and Trilipix) - Patients with disturbances of lipid metabolism such as pathologic hyperlipidemia (including congenital hypertriglyceridemia or cholesterolemia), lipoid nephrosis, or acute pancreatitis
* Patient has uncontrolled Type 1 or 2 diabetes mellitus
* Patient has another active medical condition(s) or organ disease(s) that may either compromise patient safety or interfere with the safety and/or outcome (e.g., survival) evaluation of the study drugs
* Patient or physician plans surgical treatment of malignancy, radiation therapy, or biological treatment for cancer including immunotherapy while on study, other than surgical bypass or stent insertion for relief of bile flow blockage
* Patient has a known allergy to soybeans (used in production of Kanglaite Injection) or Job's Tear (source of active ingredient of Kanglaite Injection), or to gemcitabine
* Patient has NYHA congestive heart failure Class II or higher from any cause
* Patient has unstable angina or history of an MI within 12 months
* Patient is pregnant or lactating
* Patient has used or plans to use another investigational agent within four weeks prior to screening through the entire study period including study termination and the follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Length of study

SECONDARY OUTCOMES:
Objective Response Rate | Length of study
Survival | From randomization until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Schwartzberg, MD, Principal Investigator — The West Clinic
Locations (42):
- United States (42):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Donald W. Hill, MD, Casa Grande, Arizona
  - East Valley Hematology & Oncology Medical Group, Burbank, California
  - The Oncology Institute of Hope and Innovation, Downey, California
  - Cancer Care Associates of Fresno Medical Group (California Cancer Care), Fresno, California
  - Loma Linda Oncology Medical Group, Inc., Redlands, California
  - Cancer Prevention and Treatment Center, Soquel, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Tampa General Hospital, Tampa, Florida
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Hematology / Oncology of the North Shore, Skokie, Illinois
  - Hematology Oncology of Indiana, Indianapolis, Indiana
  - McFarland Clinic, Ames, Iowa
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Research Medical Center, Kansas City, Missouri
  - Southeast Nebraska Hematology & Oncology Consultants, Lincoln, Nebraska
  - Las Vegas Cancer Center, Henderson, Nevada
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - Regional Cancer Care Associates, Howell Township, New Jersey
  - Atlantic Hematology Oncology Associates, Manasquam, New Jersey
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Arena Oncology Associates, Lake Success, New York
  - Morton Coleman, MD, New York, New York
  - Abraham Mittelman, MD, Purchase, New York
  - Richmond University Medical Center, Staten Island, New York
  - Bruckner Oncology, The Bronx, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Promedica Cancer Institute, Sylvania, Ohio
  - Hematology and Oncology Associates of NE PA, Dunmore, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Assoc, Lemoyne, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Oncology Consultants PA, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - St. Luke's Cancer Center, Houston, Texas
  - Blood And Cancer Center of East Texas, Tyler, Texas
  - Tyler Hematology Oncology, Tyler, Texas
  - Providence Regional Cancer Partnership, Everett, Washington

REFERENCES:
- [Derived] Schwartzberg LS, Arena FP, Bienvenu BJ, Kaplan EH, Camacho LH, Campos LT, Waymack JP, Tagliaferri MA, Chen MM, Li D. A Randomized, Open-Label, Safety and Exploratory Efficacy Study of Kanglaite Injection (KLTi) plus Gemcitabine versus Gemcitabine in Patients with Advanced Pancreatic Cancer. J Cancer. 2017 Jul 3;8(10):1872-1883. doi: 10.7150/jca.15407. eCollection 2017. PMID 28819385